CLINICAL TRIAL: NCT03191253
Title: Changing Health Through Food Support (CHEFS): Pilot RCT to Identify Potential Health Impacts of Providing Comprehensive, Medically-appropriate Food Support to Low-income Urban Adults Living With HIV (PLHIV)
Brief Title: Changing Health Through Food Support (CHEFS) Program
Acronym: CHEFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Project Open Hand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P0515916
Record Dates: First submitted 2017-06-07; First posted 2017-06-19 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: HIV/AIDS
Keywords: food insecurity; community-based; food assistance; food support; intervention; medically tailored; nutrition
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: We will randomize 200 participants to the intervention (n=100) or control (n=100). The intervention consists of providing comprehensive, medically-appropriate food support, individual nutritional counseling, and group-based nutritional education over 6 months to low-income clients who have been diagnosed with HIV in order to improve their viral load and health-related quality of life (primary outcomes) as well as depression, ART adherence, food security and diet quality (secondary outcomes).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention consists of comprehensive, medically-appropriate food support (meals and groceries), individual nutritional counseling, and group-based nutritional education.
  Interventions: Other: Medically-appropriate meals and groceries
- Control (No Intervention): The control group will continue to receive their regular Project Open Hand services (standard of care) which includes 1-2 food services/day.

INTERVENTIONS:
Other: Medically-appropriate meals and groceries — Full nutrition Intervention Components: (1) 7 pre-packaged frozen meals; (2) Groceries or another 7-pack of meals; (3) Nutritional supplement bag to round out the nutrition in terms of nutrients, or dietary reference intakes (DRIs), and number of servings from fruits/vegetables, whole grains, legumes, nuts/seeds and dairy. The nutritional supplemental bag will also contain bulk ingredients to aid in cooking e.g., cooking oil, spices, and herbs as well as bulk items e.g., jar of peanut butter, quart of milk; (4) Individual nutritional counseling (x2 sessions); and (5) Group nutrition education classes (X3 classes) by POH registered dietitian (RD) team.
  Arms: Intervention

SUMMARY:
UCSF and Project Open Hand (POH), a community based organization in San Francisco which provides meals and groceries to chronically ill clients in the Bay Area, have partnered to conduct an initial randomized controlled trial (RCT) of the Changing Health through Food Support (CHEFS) pilot intervention implemented by POH. The intervention consists of providing comprehensive, medically-appropriate food support, individual nutritional counseling, and group-based nutritional education over 6 months to low-income clients who have been diagnosed with HIV in order to improve their viral load and health-related quality of life (primary outcomes) as well as depression, ART adherence, food security and diet quality (secondary outcomes). We will randomize 200 participants to the intervention (n=100) or control (n=100). Participants will be followed for 6 months. The investigators will assess outcomes at baseline and 6-month follow-up using a quantitative survey and blood draws. In addition, the investigators will conduct a qualitative study at follow-up in a subset of participants to understand perceived impacts, barriers and facilitators.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* Income at or below 200% FPL (~$2400/month)
* 30-50% minimum POH regular program adherence level (i.e. regular service access rate)
* Are willing and able to eat food from POH based on one of POH's regularly available diet choices (including regular, non-dairy, vegetarian, vegetarian non-dairy, diabetic, and bland), excluding the renal diet.
* Have access to a refrigerator or freezer with sufficient space to store perishable food provided by POH, and have access to an appliance to reheat food.

Exclusion Criteria:

* Do not speak Spanish or English
* Do not have adequate cognitive or hearing capacity to complete interviews
* Have a history of violent behavior at POH (such as verbal or physical abuse to other clients and/or staff)
* Have renal disease requiring a special renal diet
* Have severe food allergies
* Currently pregnant or <6 months post-partum
* Unable to complete an interview due to a health condition
* Unable or unwilling to eat food from POH (based on one of POH's regularly available diet choices)
* Among people who share a household (such as partners, family members, or roommates), only one may be involved in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 191 (Actual)
Dates: Start 2016-07-06 (Actual); Primary Completion 2017-09-28 (Actual); Study Completion 2017-09-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline HIV viral load suppression at 6 months in the intervention compared to the control group | Assessed at baseline and 6 months
  Nondetectable HIV viral load
Change from baseline health-related quality of life at 6 months in the intervention compared to the control group | Assessed at baseline and 6 months
  Short-form SF-36, a validated tool to assess health-related quality of life

SECONDARY OUTCOMES:
Change from baseline depression at 6 months in the intervention compared to the control group | Assessed at baseline and 6 months
  Patient Health Questionnaire (PHQ-9), a validated tool to diagnose the severity of depression
Change from baseline ART adherence at 6 months in the intervention compared to the control group | Assessed at baseline and 6 months
  Visual Analogue Scale (VAS), a measure of adherence validated among people living with HIV
Change from baseline diet quality at 6 months in the intervention compared to the control group | Assessed at baseline and 6 months
  18-items adapted from National Cancer Institute Multifactor Screener, a validated tool to assess approximate intakes of fruits, vegetables, fats, proteins, dairy, grains, and sugars
Change from baseline food security at 6 months in the intervention compared to the control group | Assessed at baseline and 6 months
  U.S. Household Food Security Survey (HFSS), a validated tool to assess food insecurity

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data.

REFERENCES:
- [Background] Palar K, Napoles T, Hufstedler LL, Seligman H, Hecht FM, Madsen K, Ryle M, Pitchford S, Frongillo EA, Weiser SD. Comprehensive and Medically Appropriate Food Support Is Associated with Improved HIV and Diabetes Health. J Urban Health. 2017 Feb;94(1):87-99. doi: 10.1007/s11524-016-0129-7. PMID 28097614
- [Background] Whittle HJ, Palar K, Seligman HK, Napoles T, Frongillo EA, Weiser SD. How food insecurity contributes to poor HIV health outcomes: Qualitative evidence from the San Francisco Bay Area. Soc Sci Med. 2016 Dec;170:228-236. doi: 10.1016/j.socscimed.2016.09.040. Epub 2016 Oct 19. PMID 27771206
- [Background] Weiser SD, Hatcher AM, Hufstedler LL, Weke E, Dworkin SL, Bukusi EA, Burger RL, Kodish S, Grede N, Butler LM, Cohen CR. Changes in Health and Antiretroviral Adherence Among HIV-Infected Adults in Kenya: Qualitative Longitudinal Findings from a Livelihood Intervention. AIDS Behav. 2017 Feb;21(2):415-427. doi: 10.1007/s10461-016-1551-2. PMID 27637497
- [Background] Palar K, Laraia B, Tsai AC, Johnson MO, Weiser SD. Food insecurity is associated with HIV, sexually transmitted infections and drug use among men in the United States. AIDS. 2016 Jun 1;30(9):1457-65. doi: 10.1097/QAD.0000000000001095. PMID 26990632
- [Background] Whittle HJ, Palar K, Napoles T, Hufstedler LL, Ching I, Hecht FM, Frongillo EA, Weiser SD. Experiences with food insecurity and risky sex among low-income people living with HIV/AIDS in a resource-rich setting. J Int AIDS Soc. 2015 Nov 4;18(1):20293. doi: 10.7448/IAS.18.1.20293. eCollection 2015. PMID 26546789
- [Background] Whittle HJ, Palar K, Hufstedler LL, Seligman HK, Frongillo EA, Weiser SD. Food insecurity, chronic illness, and gentrification in the San Francisco Bay Area: An example of structural violence in United States public policy. Soc Sci Med. 2015 Oct;143:154-61. doi: 10.1016/j.socscimed.2015.08.027. Epub 2015 Aug 20. PMID 26356827
- [Background] Singer AW, Weiser SD, McCoy SI. Does Food Insecurity Undermine Adherence to Antiretroviral Therapy? A Systematic Review. AIDS Behav. 2015 Aug;19(8):1510-26. doi: 10.1007/s10461-014-0873-1. PMID 25096896
- [Background] Vogenthaler NS, Kushel MB, Hadley C, Frongillo EA Jr, Riley ED, Bangsberg DR, Weiser SD. Food insecurity and risky sexual behaviors among homeless and marginally housed HIV-infected individuals in San Francisco. AIDS Behav. 2013 Jun;17(5):1688-93. doi: 10.1007/s10461-012-0355-2. PMID 23086429
- [Background] Weiser SD, Young SL, Cohen CR, Kushel MB, Tsai AC, Tien PC, Hatcher AM, Frongillo EA, Bangsberg DR. Conceptual framework for understanding the bidirectional links between food insecurity and HIV/AIDS. Am J Clin Nutr. 2011 Dec;94(6):1729S-1739S. doi: 10.3945/ajcn.111.012070. Epub 2011 Nov 16. PMID 22089434
- [Derived] Palar K, Sheira LA, Frongillo EA, O'Donnell AA, Napoles TM, Ryle M, Pitchford S, Madsen K, Phillips B, Riley ED, Weiser SD. Food Is Medicine for Human Immunodeficiency Virus: Improved Health and Hospitalizations in the Changing Health Through Food Support (CHEFS-HIV) Pragmatic Randomized Trial. J Infect Dis. 2025 Mar 17;231(3):573-582. doi: 10.1093/infdis/jiae195. PMID 38696724